CLINICAL TRIAL: NCT06442371
Title: Additional Effects of Quranic Listening Meditation in Combination With High Intensity Interval Training on Cardiovascular Fitness and Mental Health in Obese Adults
Brief Title: Additional Effects of Quranic Listening Meditation in Combination With High Intensity Interval Training in Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Rec/01809 Warda Zaman
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity interval training + Quranic Listening (Experimental)
  Interventions: Other: High Intensity interval training + Quranic Listening
- High Intensity interval training (Active Comparator)
  Interventions: Other: High intensity interval training

INTERVENTIONS:
Other: High Intensity interval training + Quranic Listening — In this group, participants will receive protocol of High Intensity interval training which includes squats, jumping jacks, front kicks and rope jumps 3 days per week for 6 weeks, including warmup and cool down session along with Quranic listening meditation.
  Arms: High Intensity interval training + Quranic Listening
Other: High intensity interval training — In this group, participants will receive only High intensity interval training which includes squats, jumping jacks, front kicks and rope jumps 3 days per week for 6 weeks, including warmup and cool down periods with no Quranic listening meditation
  Arms: High Intensity interval training

SUMMARY:
To determine the additional effects of Quranic listening meditation, in combination with High-Intensity Interval Training on cardiovascular fitness and mental health in obese adults.

ELIGIBILITY:
Inclusion Criteria:

* Obese adults (BMI ≥ 30)
* Age range: 18-45 years
* No previous experience with Quranic listening meditation since last 4 weeks.
* No contraindications for engaging in high-intensity physical activity
* Able to attend regular sessions at clinic and follow the study protocol.
* Willingness to undergo pre and post-assessments for cardiovascular fitness and mental health measures.

Exclusion Criteria:

* Individuals with a history of the medical condition being studied
* Those who are currently taking medication that may affect the study
* Participants with a history of mental health disorders
* Individuals who are pregnant or breastfeeding
* Those who have previously participated in a similar study
* Participants with a history of substance abuse or addiction

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Modified BORG Scale | 6 week
  The Modified Borg Dyspnea Scale is numerical rating scale ranging from 0 to 10 and is used to measure dyspnea that patient report during sub-maximal exercise and is regularly administered during six-minute walk test. Changes from the baseline will be measured
6 Min walk test (Distance in meters) | 6 week
  Changes from the baseline, Body Mass Index can be define as statistical index utilizing an individual's height and weight to give an estimation of muscle versus fat in female and male of all ages. It is determined by taking an individual weight in kilograms, separated by their height in meters squared, or BMI = weight (in kg)/height (in m square).
Peak VO2 with formula | 6 week
  A generalized equation can be used to determined peak VO2 (Peak rate of oxygen consumption). The generalized equation can be used to accurately estimate mean peak VO2 from mean 6 MWD, among groups of patients with diverse diseases without the need for cardiopulmonary exercise testing. The equation is:
  Mean peak VO2(ml/kg/mins) = 4.948 + 0.023*Mean 6 MWD (meter) Changes From the Baseline will be measured
Body Mas Index | 6 week
  Changes from the baseline, Body Mass Index can be define as statistical index utilizing an individuals height and weight to give an estimation of muscle versus fat in female and male of all ages. It is determined by taking an individual weight in kilograms, separated by their height in meters squared, or BMI = weight (in kg)/height (in m square).
Heart Rate recovery | 6 week
  Heart rate recovery (HRR) is a measurement of how quickly your heart can settle back into its normal state following a workout. It is the variation in heart rate between the time when you are exercising and when you stop.
Depression Anxiety and Stress Scale | 6 week
  Depression Anxiety and Stress Scale DASS (-42), The 42-item DASS-42 self-report scale was designed to measure the negative emotional states of stress, anxiety, and depression. As part of the larger process of clinical assessment, the DASS's main value in a clinical environment is to identify the location of emotional disturbance. The DASS's primary purpose is to evaluate the severity of the main symptoms of stress, anxiety, and depression.
Systolic and diastolic blood pressure | 6 week
  Changes from the Baseline, Systolic Blood pressure (SBP) and Diastolic Blood Pressure (DBP) will be measured through sphygmomanometer
Change in blood lipid profile | 6 week
  Change in plasma total cholesterol, high density lipoproteins cholesterol (HDL), and low density lipoproteins cholesterol (LDL) after each treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, PhD*, Principal Investigator — Riphah International University
Locations (1):
- physiotherapy department, Jinnah international hospital, Abbottābād, Khyber PkahtoonKhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No